CLINICAL TRIAL: NCT04954482
Title: Anatomical and Biomechanical Study of Combined Reconstruction in the Treatment of III° Posterior Cruciate Ligament Injury
Brief Title: Anatomical and Biomechanical Study of Combined Reconstruction in III° Posterior Cruciate Ligament Injury
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liu Ping, chief physician, Peking University Third Hospital
Other Study IDs: M2017121
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Posterior Cruciate Ligament Tear
Keywords: posterior cruciate ligament; biomechanics; Combined reconstruction technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The experimental group: The included specimens were used to establish a new posterior fork reconstruction procedure.
  Interventions: Other: No Intervention
- The validation group: The included specimens were used to validate the new posterior fork reconstruction procedure.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observation study, with no intervention

SUMMARY:
To establish a III°PCL injury model on fresh cadaver knee specimens, and to define the pathological and anatomical connotation of III°PCL injury by using anatomical methods.

To explore and establish combined reconstruction techniques, including PCL reconstruction combined with injury repair and reconstruction, and to explore the role of combined reconstruction techniques in maintaining knee stability through biomechanical experiments.

DETAILED DESCRIPTION:
Objective: (1) To establish a III°PCL injury model on fresh cadaver knee specimens, and to define the pathological and anatomical connotation of III°PCL injury by using anatomical methods.

(2) To explore and establish combined reconstruction techniques, including PCL reconstruction combined with injury repair and reconstruction, and to explore the role of combined reconstruction techniques in maintaining knee stability through biomechanical experiments.

Design: ① The subjects of this study were fresh cadaver knee specimens.

* Sample size:

A Anatomical study of injury model, planning 6 cases. B. Exploration of treatment methods for complicated injuries. 8 cases of specimens are planned to be used. According to the pathological and anatomical content of III°PCL injury (IKDC standard), the repair and reconstruction techniques of combined injury were designed. Arthroscopic transtibial single-bundle PCL reconstruction technique was used in all the reconstruction of PCL. Using the robotic arm or universal sensor test system as the biomechanical test platform, Biomechanical tests were carried out on the experimental specimens, and the results were compared to determine the shortcomings of the new PCL reconstruction, according to which the surgical procedures were improved, and then the biomechanical tests were carried out. After repeated technical improvement (4 cycles, 2 specimens per cycle), the new PCL reconstruction technique was finally determined.

C To investigate the effect of new PCL reconstruction in maintaining the stability of knee joint, 8 cases were treated with a specimen plan. Biomechanical tests were performed on each specimen in its intact state, post-traumatic state (after the establishment of the III°PCL injury model), and post-traumatic state (after the application of the new PCL reconstruction technology) using the robotic arm/universal sensor test system.

Outcome evaluation: The biomechanical characteristics of knee specimens under different conditions were measured, compared and statistically analyzed, and the conclusions were drawn.

Statistical Methods:

* Multivariate linear analysis model and Bonferroni multiple comparison were used to compare the kinematics changes of knee joints under various loading conditions and knee flexion angles under the condition of knee joint integrity, III°PCL injury, PCL reconstruction, and combined injury treatment.

  * Univariate repeated measure ANOVA was used to compare the knee joint integrity, III°PCL injury, the stability of the knee joint after PCL reconstruction, and the stability of the knee joint after combined injury treatment (including the back drawer test and stress radiograph measurement).

ELIGIBILITY:
Inclusion Criteria:

• no sports injuries such as knee ligament rupture and meniscus injury specimens

Exclusion Criteria:

• sports injuries such as knee ligament rupture and meniscus injury specimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There were no sports injuries such as knee ligament rupture and meniscus injury.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
The distance of posterior displacement of the tibia | On the day of enrollment.
  The robotic arm/universal sensor test system was used as the test platform to test the specimens .

SECONDARY OUTCOMES:
Internal rotation angle of the tibia | On the day of enrollment.
  The robotic arm/universal sensor test system was used as the test platform to test the specimens .
External rotation angle of the tibia | On the day of enrollment.
  The robotic arm/universal sensor test system was used as the test platform to test the specimens .
Tibia varus Angle | On the day of enrollment.
  The robotic arm/universal sensor test system was used as the test platform to test the specimens .
Tibial valgus Angle | On the day of enrollment.
  The robotic arm/universal sensor test system was used as the test platform to test the specimens .

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No